CLINICAL TRIAL: NCT03717948
Title: Examining the Impact of Acute Blood Flow Restricted Aerobic Exercise on PGC-1α mRNA Expression in Young Healthy Males: A Randomized Cross-over Trial
Brief Title: Examining the Impact of Blood Flow Restricted Aerobic Exercise on PGC-1α mRNA Expression in Young Healthy Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Brendon Gurd, Associate Professor, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BFRNP; 402635 (Other Grant/Funding Number: NSERC)
Record Dates: First submitted 2018-10-19; First posted 2018-10-24 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Mitochondrial Biogenesis
Keywords: Acute Exercise; Mitochondria; Skeletal Muscle; PGC1α; Mitochondrial Biogenesis; Intracellular Signalling
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation concealment, assessor blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTL - BFR (Experimental): CTL Exercise then BFR Exercise
  Interventions: Other: BFR Exercise; Other: CTL Exercise
- BFR - CTL (Experimental): BFR Exercise then CTL Exercise
  Interventions: Other: BFR Exercise; Other: CTL Exercise

INTERVENTIONS:
Other: BFR Exercise — Participants will exercise on a recumbent bike placed on a 45 degree incline (BFR).
Other: CTL Exercise — Participants will exercise on a recumbent bike placed on flat ground (CTL).

SUMMARY:
This crossover study investigates the effects of restricting arterial blood flow during cycling exercise on PGC-1α and its upstream signalling pathways. In a randomized order, participants will exercise once for 30 minutes with restricted blood flow and then will exercise once for 30 minutes with no blood flow restriction.

ELIGIBILITY:
Inclusion Criteria:

* 3 hours of physical activity per week
* No previous cycling training
* No concurrent involvement in another training program
* Body mass index < 30 kg/m2

Exclusion Criteria:

* Presence of cardiovascular disease
* Presence of metabolic disease
* Taking regular oral medication
* Current smoker

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α) messenger ribonucleic acid (mRNA) | 15 minutes before exercise and 3 hours post-exercise for both exercise sessions
  Fold-change in PGC-1α mRNA expression

SECONDARY OUTCOMES:
Catecholamine concentrations | 15 minutes before exercise and immediately post-exercise for both exercise sessions
  Catecholamine concentrations in venous blood
Total and phosphorylated p38 mitogen-activated protein kinase (MAPK) | 15 minutes before exercise and immediately post-exercise for both exercise sessions
  Fold change in p38 MAPK phosphorylation
Total and phosphorylated acetyl coenzyme A carboxylase (ACC) | 15 minutes before exercise and immediately post-exercise for both exercise sessions
  Fold change in ACC phosphorylation
Total and phosphorylated protein kinase A (PKA) | 15 minutes before exercise and immediately post-exercise for both exercise sessions
  Fold change in PKA phosphorylation
Acetylated p53 | 15 minutes before exercise and immediately post-exercise for both exercise sessions
  Fold change in acetylated p53
Blood lactate | During both exercise sessions (lactate); 15 minutes before and immediately after both exercise sessions
  Average [lactate] between conditions
Heart rate (HR) | During both exercise sessions
  Average HR between conditions
Revolutions per minute (RPM) | During both exercise sessions
  Average RPM between conditions
Ratings of perceived exertion (RPE) | During both exercise sessions
  Average RPE between conditions
Oxygenated and deoxygenated hemoglobin | During both exercise sessions and up to 10 minutes after (for cuff occlusion)
  Average oxygenated and deoxygenated hemoglobin as a percentage of same day max values

CONTACTS AND LOCATIONS:
Overall Officials: Brendon J Gurd, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT03717948/SAP_001.pdf